CLINICAL TRIAL: NCT06682195
Title: Neoadjuvant Chemotherapy Combined With Toripalimab for Triple-negative Breast Cancer : a Prospective, Single-arm, Multi-center Study (NEOTORCH-BREAST02)
Brief Title: Neoadjuvant Chemotherapy Combined With Toripalimab for TNBC (NEOTORCH-BREAST02)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20240127C-R2
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: TNBC, Triple Negative Breast Cancer
Keywords: Triple negative breast cancer; Toripalimab; Adjuvant Treatment
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant chemotherapy combined with Toripalimab (Experimental): 1, Neoadjuvant Chemotherapy Phase Combined with Toripalimab
  1. First Phase of Neoadjuvant Chemotherapy: Epirubicin + Cyclophosphamide + Toripalimab. Administered intravenously: 100 mg/m² Epirubicin + 600 mg/m² Cyclophosphamide + 240 mg Toripalimab, every 3 weeks for a total of 6 weeks.
  2. Second Phase of Neoadjuvant Chemotherapy: Albumin-bound Paclitaxel + Toripalimab. Administered intravenously: 260 mg/m² Albumin-bound Paclitaxel + 240 mg Toripalimab, every 3 weeks for a total of 6 weeks.
  2, Receive Breast Cancer Radical Surgery After 4 Cycles of Neoadjuvant Chemotherapy 3, Postoperative Adjuvant Therapy
  1. If pathology indicates pCR: Continue immunotherapy, administering 240 mg Toripalimab intravenously every 3 weeks for a total of 1 year.
  2. If pathology indicates non-PCR: Continue postoperative adjuvant chemotherapy combined with Toripalimab.
  4, Perform Gene Testing on Biopsy Tissue Before Treatment, and Collect Blood Samples for ctDNA Testing Before and After Treatment.
  Interventions: Drug: Neoadjuvant chemotherapy combined with Toripalimab

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy combined with Toripalimab — 1, Neoadjuvant Chemotherapy Phase Combined with Toripalimab
  1. First Phase of Neoadjuvant Chemotherapy: Epirubicin + Cyclophosphamide + Toripalimab. Administered intravenously: 100 mg/m² Epirubicin + 600 mg/m² Cyclophosphamide + 240 mg Toripalimab, every 3 weeks for a total of 6 weeks.
  2. Second Phase of Neoadjuvant Chemotherapy: Albumin-bound Paclitaxel + Toripalimab. Administered intravenously: 260 mg/m² Albumin-bound Paclitaxel + 240 mg Toripalimab, every 3 weeks for a total of 6 weeks.
  2, Receive Breast Cancer Radical Surgery After 4 Cycles of Neoadjuvant Chemotherapy 3, Postoperative Adjuvant Therapy
  1. If pathology indicates pCR: Continue immunotherapy, administering 240 mg Toripalimab intravenously every 3 weeks for a total of 1 year.
  2. If pathology indicates non-PCR: Continue postoperative adjuvant chemotherapy combined with Toripalimab.
  4, Perform Gene Testing on Biopsy Tissue Before Treatment, and Collect Blood Samples for ctDNA Testing Before and After Treatment.

SUMMARY:
This study is a prospective, single arm, multi-center phase II clinical trial. The primary study objective is to evaluate the pathologic complete response（PCR） of Adjuvant treatment of TNBC breast cancer with Toripalimab combined with neoadjuvant chemotherapy, including the incidences and types of adverse events. The secondary study objective is to observe and evaluate the disease-free survival (DFS), Progression-Free-Survival (PFS ),and Objective Response Rate(ORR)

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-70 years old;
2. ECOG score is 0-1 points;
3. Histologically proven tumors >1cm in diameter (T1c-3; N0-2; M0) invasive breast cancer;
4. All patients had triple negative breast cancer confirmed by histopathology;
5. Pathological examination of PD-L1 expression:

   The Combined Positive Score (CPS) refers to the percentage of PD-L1 positive cells (including tumor cells, lymphocytes, macrophages) in all tumor cells. Our center detected the PD-L1 antibody site as 22C3.
6. The functional level of major organs must meet requirements
7. For female patients who have not yet reached menopause or undergone surgical sterilization: during the treatment period and in the study treatment, the final use effective contraceptive methods for at least 6 months after a single administration.
8. Voluntarily join this study, sign an informed consent form, have good compliance, and are willing to cooperate with follow-up.

Exclusion Criteria:

1. Stage IV breast cancer.
2. Inflammatory breast cancer.
3. Previously received anti-tumor treatment or radiation therapy for any malignant tumor, excluding those that have been cured Malignant tumors such as cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma.
4. Simultaneously undergoing anti-tumor treatment in other clinical trials, including but not limited to chemotherapy and endocrine therapy. Treatment, biological therapy, bone improvement drug therapy, or immune checkpoint inhibitor therapy, etc.
5. The patient had undergone major surgical procedures unrelated to breast cancer within 4 weeks before the first administration of the study drug, or the patient has not fully recovered from such surgical procedures.
6. Serious heart disease or discomfort, including but not limited to the following diseases:

1) Diagnosed history of heart failure or systolic dysfunction (LVEF less than 50%).2) High risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate greater than 100bpm, significant ventricular arrhythmias (such as ventricular tachycardia), or higher-level atrioventricular block (i.e. Mobitz II second or third degree atrioventricular block).3) Angina requiring medication for treatment. 4) Heart valve disease with clinical significance. 5) ECG shows transmural myocardial infarction. 6) Poor control of hypertension (systolic blood pressure greater than 180mmHg and/or diastolic blood pressure greater than 180mmHg after drug treatment) 100mmHg).

7. Uncontrolled active infections that require treatment; History of immunodeficiency, including HIV testing positive Sexual, or suffering from other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation.

8. Patients with chronic active hepatitis B or active hepatitis C (excluding hepatitis B virus carriers, stable hepatitis B after drug treatment [HBV-DNA test negative or<50IU/ml] and cured hepatitis C patients [HCV RNA test negative]).

9. Have received immunotherapy and experienced adverse immune events such as immune related pneumonia and myocarditis, which have been determined by researchers to potentially affect the safety of the experimental medication.

10. Individuals with a known history of allergies to the components of this medication regimen.

11. Pregnant and lactating female patients, female patients with fertility and positive baseline pregnancy test results, or reproductive age patients who are unwilling to take effective contraceptive measures during the entire trial period and within 6 months after the last study medication.

12. Suffering from serious accompanying diseases or other comorbidities that may interfere with the planned treatment, or any other circumstances that the researcher deems unsuitable for the patient to participate in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response（PCR） | 2 years
  The primary study objective is to evaluate the pathologic complete response（PCR） of Neodjuvant treatment of TNBC breast cancer with Toripalimab combined with neoadjuvant chemotherapy and sequential Toripalimab monoclonal antibody

SECONDARY OUTCOMES:
Event-free survival (EFS) | 3 years
radiologic complete response (rCR) | 3 years
Objective Response Rate(ORR) | 3 years

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Nanchang People's Hospital, Nanchang, Jiangxi
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou
  - The First Affiliated Hospital of Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Jinhua Municipal Central Hospital, Jinhua
  - Nantong First People's Hospital, Nantong
  - Zhongshan Hospital, Fudan University, Shanghai
  - Shanxi Provincial Cancer Hospital, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xinjiang Medical University Affiliated Cancer Hospital, Xinjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou